CLINICAL TRIAL: NCT03556137
Title: Use of [18F]FTC-146 PET/MRI in the Diagnosis of Chronic Pain
Brief Title: PET/MRI in the Diagnosis of Chronic Pain
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Anand Veeravagu, Assistant Professor of Neurosurgery, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 45332
Record Dates: First submitted 2018-06-02; First posted 2018-06-14 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Neuropathic Pain; Nociceptive Pain; Mixed Pain (Nociceptive and Neuropathic); Spinal Pain; Radiculopathy; Myelopathy; Neurogenic Claudication
Keywords: PET/MRI; Chronic Pain
MeSH Terms: conditions — Neuralgia; Nociceptive Pain; Radiculopathy; Spinal Cord Diseases; Chronic Pain | interventions — 6-(3-fluoropropyl)-3-(2-(azepan-1-yl)ethyl)benzo(d)thiazol-2(3H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pain Patients (Experimental): Individuals suffering from nociceptive pain, neuropathic pain, and mixed pain (pain that appears to be both nociceptive and neuropathic) and undergo a [18F]FTC-146 PET/MRI scan.
  Interventions: Drug: [18F]FTC-146
- Healthy Volunteers (Experimental): Individuals who do not have pain and undergo a [18F]FTC-146 PET/MRI scan.
  Interventions: Drug: [18F]FTC-146

INTERVENTIONS:
Drug: [18F]FTC-146 — Adult participants will be injected with 5-10 mCi of [18F]FTC-146 and undergo a PET/MRI scan.
  Other Names: S1R

SUMMARY:
Several studies have implicated involvement of sigma-1 receptors (SR1s) in the generation of chronic pain, while others are investigating anti SR1 drugs for treatment of chronic pain. Using [18F]-FTC-146 and positron emission tomography/magnetic resonance imaging (PET/MRI), the investigators hope to identify the source of pain generation in patients with chronic pain. The purpose of this study is to compare the uptake of [18F]FTC-146 in healthy volunteers to that of individuals suffering from chronic pain.

DETAILED DESCRIPTION:
Chronic pain is a significant, widespread problem affecting every fifth person worldwide. Reported in 2011 by the Institute of Medicine, chronic pain affects 116 million American adults - more than the total number of individuals affected by heart disease, cancer, and diabetes combined. An estimated $635 billion each year is spent in the medical management of chronic pain and lost productivity. Better clinical methods to diagnose and localize pain are needed.

The investigators have developed a S1R-specific radiotracer, [18F]FTC-146. Using imaging approaches to assess the location of S1R in pain may provide a tool to diagnose pain generators, monitor treatment response, and aid in the selection of patients for treatment.

The goal is to use [18F]FTC-146 to image S1R expression in healthy volunteers and to compare the images to those individuals suffering from pain conditions in the following categories: (1) nociceptive pain (pain that results from tissue injury or inflammation), (2) neuropathic pain (pain that results from direct injury, disruption, impingement/compression or malfunction of the peripheral and/or central nervous system), and (3) mixed pain (pain that appears to have both nociceptive and neuropathic).

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

1. At least 18 years old.
2. Covid Vaccination status: Vaccinated or unvaccinated subjects who received a negative test result from the Covid test within 72 hours of the scan.

Pain Patients:

1. At least 18 years old.
2. Chronic pain (nociceptive, neuropathic or mixed pain) lasting greater than 2 months.
3. Pain level of at least 4/10 on a 0-10 Comparative Pain Scale.
4. Covid Vaccination status: Vaccinated or unvaccinated subjects who received a negative test result from the Covid test within 72 hours of the scan.

Exclusion Criteria:

Healthy Volunteers:

1. Pain
2. Pain Medication
3. MRI incompatible
4. Pregnant or nursing
5. Non-English speaker
6. Claustrophobic

Pain Patients:

1. MRI incompatible
2. Pregnant or nursing
3. Non-English speaker
4. Claustrophobic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
[18F]FTC-146 Biodistribution in Healthy Volunteers | Estimated average of 3 hours
  Biodistribution of [18F]FTC-146 represented as Standardized Uptake Value max (SUVmax) in healthy volunteers.
[18F]FTC-146 Biodistribution in Pain Patients | Estimated average of 3 hours
  Biodistribution of [18F]FTC-146 represented as Standardized Uptake Value max (SUVmax) in pain patients.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Veeravagu, MD, Principal Investigator — Stanford University Department of Neurosurgery
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shen B, Behera D, James ML, Reyes ST, Andrews L, Cipriano PW, Klukinov M, Lutz AB, Mavlyutov T, Rosenberg J, Ruoho AE, McCurdy CR, Gambhir SS, Yeomans DC, Biswal S, Chin FT. Visualizing Nerve Injury in a Neuropathic Pain Model with [18F]FTC-146 PET/MRI. Theranostics. 2017 Jul 8;7(11):2794-2805. doi: 10.7150/thno.19378. eCollection 2017. PMID 28824716
- [Background] Hjornevik T, Cipriano PW, Shen B, Park JH, Gulaka P, Holley D, Gandhi H, Yoon D, Mittra ES, Zaharchuk G, Gambhir SS, McCurdy CR, Chin FT, Biswal S. Biodistribution and Radiation Dosimetry of 18F-FTC-146 in Humans. J Nucl Med. 2017 Dec;58(12):2004-2009. doi: 10.2967/jnumed.117.192641. Epub 2017 Jun 1. PMID 28572487
- [Background] Shen B, Park JH, Hjornevik T, Cipriano PW, Yoon D, Gulaka PK, Holly D, Behera D, Avery BA, Gambhir SS, McCurdy CR, Biswal S, Chin FT. Radiosynthesis and First-In-Human PET/MRI Evaluation with Clinical-Grade [18F]FTC-146. Mol Imaging Biol. 2017 Oct;19(5):779-786. doi: 10.1007/s11307-017-1064-z. PMID 28280965
- [Background] Shen B, James ML, Andrews L, Lau C, Chen S, Palner M, Miao Z, Arksey NC, Shuhendler AJ, Scatliffe S, Kaneshige K, Parsons SM, McCurdy CR, Salehi A, Gambhir SS, Chin FT. Further validation to support clinical translation of [(18)F]FTC-146 for imaging sigma-1 receptors. EJNMMI Res. 2015 Dec;5(1):49. doi: 10.1186/s13550-015-0122-2. Epub 2015 Sep 17. PMID 26384292
- [Background] James ML, Shen B, Nielsen CH, Behera D, Buckmaster CL, Mesangeau C, Zavaleta C, Vuppala PK, Jamalapuram S, Avery BA, Lyons DM, McCurdy CR, Biswal S, Gambhir SS, Chin FT. Evaluation of sigma-1 receptor radioligand 18F-FTC-146 in rats and squirrel monkeys using PET. J Nucl Med. 2014 Jan;55(1):147-53. doi: 10.2967/jnumed.113.120261. Epub 2013 Dec 12. PMID 24337599
- [Derived] Yoon D, Fast AM, Cipriano P, Shen B, Castillo JB, McCurdy CR, Mari Aparici C, Lum D, Biswal S. Sigma-1 Receptor Changes Observed in Chronic Pelvic Pain Patients: A Pilot PET/MRI Study. Front Pain Res (Lausanne). 2021 Oct 20;2:711748. doi: 10.3389/fpain.2021.711748. eCollection 2021. PMID 35295458